CLINICAL TRIAL: NCT02648048
Title: A Single Arm, Multicenter, Open-label, Phase 1b Study to Assess the Safety and Tolerability of Oral Vismodegib in Combination With Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Study of Oral Vismodegib in Combination With Pirfenidone in Participants With Idiopathic Pulmonary Fibrosis
Acronym: ISLAND2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB29764; 2015-003481-81 (EudraCT Number)
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Vismodegib; Pirfenidone
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone; HhAntag691

ARMS (1):
- Vismodegib and Pirfenidone (Experimental): Participants being treated with pirfenidone, will receive vismodegib 150 milligrams (mg) once daily and pirfenidone up to 2403 mg daily orally for 24 weeks.
  Interventions: Drug: Pirfenidone; Drug: Vismodegib

INTERVENTIONS:
Drug: Pirfenidone — Pirfenidone will be administered as per the dosage schedule mentioned in arm description.
  Other Names: RO0220912
Drug: Vismodegib — Vismodegib will be administered as per the dosage schedule mentioned in arm description.
  Other Names: RO5450815

SUMMARY:
This is a single arm, multicenter, open-label, Phase 1b study to evaluate the safety and tolerability of vismodegib in combination with pirfenidone in participants with idiopathic pulmonary fibrosis (IPF) currently being treated with pirfenidone.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of IPF 5 years from time of screening, confirmed at baseline
* Tolerated dose of pirfenidone 1602-2403 mg once daily (QD) for a minimum of 24 weeks required prior to and during screening
* Greater than or equal to (>=) 50 percent (%) and less than or equal to (<=) 100% of predicted forced vital capacity (FVC) at screening
* Stable baseline lung function as evidenced by a difference of less than (<) 10% in absolute FVC measurements (in liters) between screening and Day 1/Visit 2 prior to enrollment
* >=30% and <=90% of predicted diffusion capacity of the lung for carbon monoxide at screening
* Agree to use protocol defined methods of contraception
* Male participants must agree not to donate semen during the study and for at least 2 months (or as per local requirements) after the last dose of vismodegib
* Agree not to donate blood or blood products during the study and for at least 9 months (or as per local requirements) after the last dose of study treatment

Exclusion Criteria:

* Prior treatment with vismodegib or any Hh-pathway inhibitor
* Evidence of other known causes of interstitial lung disease
* Hospitalization due to an exacerbation of IPF within 4 weeks prior to or during screening
* Lung transplant expected within 6 months of screening
* Evidence of clinically significant lung disease other than IPF
* Post-bronchodilator forced expiratory volume in 1 second/FVC ratio <0.7 at screening
* Any clinically significant medical disease (other than IPF) that is associated with an expected survival of <6 months, likely to require a change in therapy during the study
* Class IV New York Heart Association chronic heart failure or historical evidence of left ventricular ejection fraction <35%
* Known current malignancy or current evaluation for a potential malignancy
* Known immunodeficiency, including, but not limited to, human immunodeficiency virus infection
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Creatinine clearance <=30 milliliter per minute, calculated using the Cockcroft-Gault formula

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious and Non-Serious Adverse Events | Baseline up to 28 weeks
  An adverse event is any untoward medical occurrence in a participant who receive study drug without regard to possibility of causal relationship. A serious adverse event is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Percentage of Participants with Discontinuation of Any Study Medication Due to a Drug-Related Adverse Event | Baseline up to 28 weeks
  An adverse event is any untoward medical occurrence in a participant who receive study drug without regard to possibility of causal relationship. Relatedness to the study drug will be assessed by the investigator.
Percentage of Participants with Dose Modifications Due to Laboratory Abnormalities and Adverse Events | Baseline up to 28 weeks
  An adverse event is any untoward medical occurrence in a participant who receive study drug without regard to possibility of causal relationship.
Percentage of Participants with Clinically Meaningful Laboratory Abnormalities as Assessed by Investigator | Baseline up to 28 weeks
  Vital signs and laboratory parameters will be evaluated, and percentage of participants with any clinically meaningful abnormalities as assessed by Investigator will be reported. Laboratory abnormalities of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade greater than (>) 3 will be considered clinical meaningful.

SECONDARY OUTCOMES:
Total and Free Trough Plasma Concentrations of Vismodegib at Week 4 (Cmin, Wk4) | Predose (0 hour) at Week 4
  Total plasma concentration of vismodegib = free (unbound) vismodegib plasma concentration + alpha-1-acid glycoprotein (AAG)-bound vismodegib plasma concentration.
Total and Free Trough Plasma Concentrations of Vismodegib at Week 12 (Cmin, Wk12) | Predose (0 hour) at Week 12
  Total plasma concentration of vismodegib = free (unbound) vismodegib plasma concentration + AAG-bound vismodegib plasma concentration.
Total and Free Trough Plasma Concentrations of Vismodegib at Week 24 (Cmin, Wk24) | Predose (0 hour) at Week 24
  Total plasma concentration of vismodegib = free (unbound) vismodegib plasma concentration + AAG-bound vismodegib plasma concentration.
Total and Free Trough Plasma Concentrations of Vismodegib at Safety Follow-up Visit (Cmin, SFU) | At Day 30 post last dose (last dose = 24 weeks) (up to 28 weeks)
  Total plasma concentration of vismodegib = free (unbound) vismodegib plasma concentration + AAG-bound vismodegib plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (14):
  - Scripps Clinic, La Jolla, California
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Suburban Lung Associates, Elk Grove, Illinois
  - Medical Consultants, PC ; Pulmonary, Muncie, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tulane University Medical School, New Orleans, Louisiana
  - Steward St. Elizabeth's Medical Center ; Pulmonary, Critical Care and Sleep Medicine, Boston, Massachusetts
  - Creighton University Medical Center, Omaha, Nebraska
  - Allied Clinical Research, Reno, Nevada
  - Atlantic Respiratory Institute, Summit, New Jersey
  - Pulmonix LLC, Greensboro, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Western Washington Medical Group, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
- Fraunhofer-Institut fur Toxikologie und Experimentelle Medizin ITEM, Hanover, Germany

REFERENCES:
- [Derived] Prasse A, Ramaswamy M, Mohan S, Pan L, Kenwright A, Neighbors M, Belloni P, LaCamera PP. A Phase 1b Study of Vismodegib with Pirfenidone in Patients with Idiopathic Pulmonary Fibrosis. Pulm Ther. 2019 Dec;5(2):151-163. doi: 10.1007/s41030-019-0096-8. Epub 2019 Jul 19. PMID 32026407